CLINICAL TRIAL: NCT03151408
Title: A Phase III, Double-Blind, Placebo-Controlled, Multicenter, Randomized Study Of Pracinostat In Combination With Azacitidine In Patients ≥18 Years With Newly Diagnosed Acute Myeloid Leukemia Unfit For Standard Induction Chemotherapy
Brief Title: An Efficacy and Safety Study Of Pracinostat In Combination With Azacitidine In Adults With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The IDMC recommended to stop the study prematurely due to a lack of efficacy.
Sponsor: Helsinn Healthcare SA (Industry)
Collaborators: Clinipace Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRAN-16-52
Record Dates: First submitted 2017-05-05; First posted 2017-05-12 (Actual); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — SB939 compound; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pracinostat plus AZA (Experimental): 60 mg capsule orally, once a day, 3 times a week for 3 weeks, followed by 1 week of rest of each 28-day cycle. As a background therapy azacitidine (AZA) will be administered at a dose of 75 mg/m2 by SC or IV injection daily for 7 days of each 28-day cycle.
  Interventions: Drug: Pracinostat; Drug: Azacitidine
- Placebo plus AZA (Placebo Comparator): 1 capsule orally, once a day, 3 times a week for 3 weeks, followed by 1 week of rest of each 28-day cycle. As a background therapy azacitidine (AZA) will be administered at a dose of 75 mg/m2 by SC or IV injection daily for 7 days of each 28-day cycle.
  Interventions: Drug: Placebos; Drug: Azacitidine

INTERVENTIONS:
Drug: Pracinostat — 60 mg capsule
  Other Names: SB939
  Arms: Pracinostat plus AZA
Drug: Placebos — capsule
  Arms: Placebo plus AZA
Drug: Azacitidine — SC or IV injection
  Other Names: AZA

SUMMARY:
This is a Phase III, multicenter, double-blind, randomized study of pracinostat vs. placebo with azacitidine (AZA) as background therapy in patients ≥ 18 years of age with newly diagnosed acute myeloid leukemia (AML), excluding acute promyelocytic leukemia and cytogenetic low-risk AML, who are unfit to receive intensive remission induction chemotherapy due to age ≥ 75 years or comorbidities. Patients will be randomized in a 1:1 ratio to one of two groups: Group A (experimental group) to receive pracinostat plus AZA and Group B (control group) to receive placebo plus AZA. Randomization will be stratified by cytogenetic risk category (intermediate vs. unfavorable-risk, according to SWOG Cytogenetic Risk Category Definitions) and ECOG performance status (0-1 vs. 2). Treatments will be administered based on 28-day cycles, with pracinostat/placebo administered orally once every other day, 3 times a week for 3 weeks, followed by one week of no treatment and AZA administered for 7 days of each cycle. Study treatment should continue until there is documented disease progression, relapse from complete remission (CR), or non-manageable toxicity. A minimum of 6 cycles may be required to achieve a complete remission. Once permanently discontinued from study treatment, patients will enter the Long-term Follow-up phase of the study and will be followed for assessment of disease progression, if applicable, and survival every 3 months (±1 month) until death. The end of this study is defined when 390 events (deaths) have occurred and the study is unblinded for final overall survival analysis. Patients who are receiving study treatment at the end of the study may have the opportunity to continue to receive the study drugs to which they were randomized to (Post- Study Observation Period), until the Sponsor informs the Investigators of the appropriate course of action based on the study results. The Post-Study Observation Period is defined as the period starting from the end of the study for a maximum of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥ 18 years of age with newly diagnosed, histologically or cytologically confirmed, AML including de novo, secondary to antecedent hematologic disorders, or treatment-related disease with intermediate or unfavorable-risk cytogenetics
2. Unable to receive intensive chemotherapy regimens at enrollment, based on one of the following:

   I. Age ≥ 75 years, or

   II. Age < 75 years with at least 1 of the following co-morbidities:
   1. An ECOG performance status of 2
   2. Clinically significant cardiovascular disease defined as:

   i. Left ventricular ejection fraction (LVEF) ≤ 50%, measured within 3 months prior to Day 1 confirmed by ECHO/MUGA ii. Congestive heart failure requiring medical therapy iii. Chronic stable angina requiring medical therapy iv. Prior cerebrovascular accident with sequelae c. Clinically significant pulmonary disease defined as: i. Forced expiratory volume in 1 second (FEV1) ≤ 65% of expected ii. Lung diffusing capacity for carbon monoxide (DLCO) ≤ 65% of expected Confirmed by pulmonary tests. d. Diabetes mellitus with symptomatic end-organ damage (e.g., retinopathy, nephropathy, neuropathy, vasculopathy) e. Autoimmune inflammatory conditions (e.g., rheumatoid arthritis, systemic lupus erythematous, inflammatory bowel disease, or similar) requiring chronic disease modifying therapy (e.g., etanercept, adalimumab, infliximab, rituximab, methotrexate, or similar) f. Class III obesity defined as a Body Mass Index (BMI) > 40 kg/m2 g. Renal impairment defined as serum creatinine > 1.3 mg/dL (> 115 µmol/L) or creatinine clearance <70 ml/min h. Clinically significant cognitive impairment defined as requiring medical therapy and/or assistance with activities of daily living
3. 20% blasts in bone marrow
4. Peripheral white blood cell (WBC) count 30,000/µL For cyto-reduction, hydroxyurea is allowed during screening and up to Cycle 1, Days 1-14, to reduce WBC count to < 30,000 µL prior to Day 1. After Cycle 1, Day 14, hydroxyurea is prohibited.
5. ECOG performance status ≤ 2
6. Adequate organ function as evidenced by the following laboratory findings:

   1. Total bilirubin ≤ 2 × upper limit of normal (ULN) or < 3 x ULN for patients with Gilbert-Meulengracht Syndrome
   2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × ULN
7. Serum creatinine ≤ 1.5 × ULN according to institutional standards or creatinine clearance ≥ 50 mL/min
8. QT-interval corrected according to Fridericia's formula (QTcF) ≤ 450 ms on electrocardiogram (ECG) at Screening
9. Male patient who is surgically sterile, or male patient who is willing to agree to remain completely abstinent (refrain from heterosexual intercourse) or who use barrier contraceptive measures and agree to refrain from donating sperm during the entire study treatment period and for 3 months after the last administration of study drug
10. Female patient who is of childbearing potential willing to use adequate contraceptive measures while participating on study, OR willing to completely abstain from heterosexual intercourse during the entire study treatment period
11. Female patient who is of childbearing potential must have a negative serum pregnancy test result within 3 weeks prior to starting study drugs.
12. Willing to provide voluntary written informed consent before performance of any study related procedure not part of normal medical care
13. Willing and able to understand the nature of this study and to comply with the study and follow-up procedures.

Exclusion Criteria:

1. Able to receive intensive induction chemotherapy
2. AML-associated inv(16)/t(16;16)/del(16q), t(15;17) (i.e. promyelocytic leukemia) with/without secondary aberrations; t(8;21) lacking del (9q) or complex karyotypes
3. Presence of an active malignant disease within the last 12 months, with the exception of adequately treated cervical cancer in-situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria]). Other malignancies may be considered after consultation with the Medical Monitor
4. Life-threatening illnesses other than AML, uncontrolled medical conditions or organ system dysfunction that, in the Investigator's opinion, could compromise the patient's safety or put the study outcomes at risk
5. Uncontrolled arrhythmias; any Class 3-4 cardiac diseases as defined by the New York Heart Association (NYHA) functional classification
6. Evidence of AML central nervous system (CNS) involvement
7. Previous chemotherapy for AML except for the following, which are allowed:

   1. Hydroxyurea for cytoreduction
   2. One course of hypomethylating agent therapy (i.e.; up to 7 doses of azacitidine or 3-5 days of decitabine) within 30 days prior to enrollment (Day 1)
8. Use of experimental drugs ≤ 30 days prior to screening
9. Received prior HDAC inhibitor therapy
10. Received prior treatment with a hypomethylating agent, except as allowed in Exclusion Criterion 7.b
11. Known hypersensitivity to any components of pracinostat, azacitidine, or mannitol
12. History of human immunodeficiency virus (HIV) or an active and uncontrolled infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
13. Gastrointestinal (GI) tract disease that causes an inability to take oral medication, malabsorption syndrome, or a requirement for IV alimentation; prior surgical procedures affecting absorption; or uncontrolled inflammatory GI disease (e.g., Crohn's disease, ulcerative colitis)
14. Any disease(s), psychiatric condition, metabolic dysfunction, or findings from a physical examination or clinical laboratory test result that would cause reasonable suspicion of a disease or condition, that contraindicates the use of pracinostat and/or AZA, that may increase the risk associated with study participation, that may affect the interpretation of the results, or that would make the patient inappropriate for this study
15. Breast-feeding woman
16. current smokers(use of patches, chewing gums and vaping nicotine conaining fluids is permitted). Patients who stopped smoking at least 8 day prior to first pracinostat dosing can be enrolled, provided they refrain from smoking during the whole study
17. prohibited concomitant medications
18. uncontrolled infections
19. receive more than 1 prior cycle of HMA or bone marrow transplant for any prior hematological disorder antecedent to AML

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2017-06-23 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2020-08-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Study Chair — MD Anderson
Locations (138):
- United States (30):
  - Mayo clinic hospital, Phoenix, Arizona
  - Arizona Oncology Associates, East Valley Cancer Center, Tempe, Arizona
  - University of Arizona cancer center-north campus, Tucson, Arizona
  - 10666 N.Torrey Pines-Scripps Cancer Center, La Jolla, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Saint alphonsus Regional medical center-cancer care center, Boise, Idaho
  - Loyola University Chicago, Maywood, Illinois
  - Universitz of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Pontchartrain Cancer Center (Research Location), Covington, Louisiana
  - Rcca Md Llc, Bethesda, Maryland
  - UMass Memorial medical center-university campus, Worcester, Massachusetts
  - Michigan Center of Medical Research, Farmington Hills, Michigan
  - Michigan State University, Lansing, Michigan
  - Mayo clinic, Rochester, Minnesota
  - Mercy Research, Springfield, Missouri
  - 100 Mercy Way, Joplin, Montana
  - Stony Brook University, Stony Brook, New York
  - Duke University Medical Center-2400 Pratt Street, Durham, North Carolina
  - University Hospital Cleveland Medical Center, Cleveland, Ohio
  - Mercy Clinic Oncology & Hematology, Oklahoma City, Oklahoma
  - Oklahoma cancer specialist and research institute, Tulsa, Oklahoma
  - GHS Cancer Institute, Greenville, South Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - VA North texas Health Care sytem,Dallas VA Medical Center div. Hematology Oncology, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Emily Couric Clinical cancer center, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - Thomas Reeve Chauncey, Seattle, Washington
- Argentina (6):
  - Hospital italiano de Buenos Aires, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - Instituto Medico Especializado Alexander Fleming, Ciudad Autonoma de Buenos Aire, Buenos Aires
  - hospital Italiano la Plata, La Plata, Buenos Aires
  - Sanatorio Britanico SA Paraguay 40, 3P, Rosario, Santa Fe Province
  - sanatorio Allende, Córdoba
  - H ospi tal Privado de Cordoba, Córdoba
- Australia (9):
  - Liverpool Hospital, Liverpool, New South Wales
  - Sunshine coast university hospital, Birtinya, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - The Northern hospital Pharmacy Department, Ground Floor, Epping, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Austin Hospital, Clinical Trial Pharmacy, Heidelberg, Victoria
  - Liverpool hospital, Liverpool
  - Royal Perth Hospital, Perth
  - Prince of Wales Hospital, Randwick
- Austria (3):
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Müllner Hauptstrabe 48, Salzburg
  - General Hospital Hietzing, Vienna
- Brazil (10):
  - Liga Paranaense de Com bate ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Ce ntro de Pesquisas Hospital Amara l Ca rvalh o, Jaú, São Paulo
  - Centro de Pesquisa Clinica do Hospital Santa Marcelina, São Paulo, São Paulo
  - Hospital de Cancer de Barretos, Barretos
  - Hospital Santa Casa de Belo Horizonte -Serviyo de Oncologia Clinica, Belo Horizonte
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis
  - Hospital de ClÃ-nicas de Porto Alegre, Porto Alegre
  - Institute Nacional de Cancer Jose de Alencar Gomes da Silva-INCA, Rio de Janeiro
  - Faculdade de Medicina do ABC - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto
- Czechia (5):
  - "Fakultni nemocnice Hradec Kralove,, Hradec Králové
  - Fakultni nemocnice Olomuc, Olomouc
  - "Fakultni nemocnice Kralovske Vinohrady,, Prague
  - Fakultni nemocnice Kralovske Vinohrady,, Prague
  - Vseobecna fakultni nemocnice, Prague
- France (7):
  - CHU Amiens Picardie-Site Sud-Service d'Hematologie, Amiens
  - L'Hopital privé du Confluent SAS, Nantes
  - CHU de Nice, Archet 1 Hospital-Hematology department, Nice
  - Hospital saints Louis, Paris
  - Haut-Leveque-Service d'hématologie clinique et de thérapie cellular, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel, Rouen
- Germany (8):
  - Klinikum St. Marien Amberg, Amberg, Bavaria
  - Universitatsklinikum Erlangen, Erlangen, Bavaria
  - Marien Hospital Herne-Universitätsklinikum der Ruhr-Universität Bochum, Herne, North Rhine-Westphalia
  - Charité-Universitätsmedizin - 1. Campus Mitte, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Staedtisches krankenhaus kiel, Kiel
  - Universitaet Mainz, Mainz
- Hungary (6):
  - university of Pécs, Pécs, Baranya
  - Pecsi Egyetem I. Belgy6gyaszati Klinika, Pécs, Baranya
  - St. Istvan & St. Laszlo Hospital, Deapartment of Hematology and Stem Cell Transplantation, Budapest
  - University of Debrecen Clinical Center, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Dep. Of Haematology, Kaposvár
  - Szabolcs-Szatmar-Bereg megyei Korhazak es Egyetemi Oktatokorhaz â€" Josa Andras Oktatokorhaz, Hematologiai Osztaly, Nyíregyháza
- Italy (13):
  - Ospedale San Raffaele-U.O. Ematologia e TMO, Milan, Lombardy
  - Ospedale la Maddalena, UO Oncoematologia e TMO, Palermo, PA
  - AOU Policlinico Consorziale di Bari, Bari
  - AOU Policlinico Sant'Orsola-Malpighi, Bologna
  - Azienda Ospedaliera-Università Careggi, Florence
  - Ospedale Policlinico San Martino, Genova
  - ospedale Vito Fazzi, Lecce
  - Azienda Ospedaliere Antonio Cardarelli,, Naples
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Fondazione IRCCS policlinico San Matteo Pavia, Pavia
  - Fondazione PTV-Policlinico Tor Vergata, Roma
  - Policlinico Universitario Gemelli, Roma
  - Azienda Ospedaliera Ordine Mauriziano, Torino
- Poland (4):
  - Wojewodzkie Wielospecjalistyczne Centrum onkologii I traumatologii, Lodz
  - Examen Sp. Z o.o.,, Poznan
  - Specjalistyc:my Szpi tal im. dra Alfreda Sokolowskiego, Wałbrzych
  - Uniwersytecki Szpital Kliniczny, Wroclaw
- Romania (6):
  - Spitalul Clinic Filantropia, Craiova, Jud.dolj
  - Spitalul Clinic Colentina, Bucharest
  - clinical hospital Coltea Bld, Bucharest
  - Spitalul Universitar de Urgenta Bucuresti, Bucharest
  - Oncological Institute "Ion Chiricuta", Cluj-Napoca
  - institutu Regional de Oncologie Iasi, Iași
- South Korea (7):
  - Inje university Busan Paik Hospital, Busan
  - Chonnam National University Hwasun Hospital, Hwasun
  - Gachon University Gil medical center, div hematology, Incheon
  - Seoul National University Hospital, Div.Hematology/Oncology, Seoul
  - Sumsung medical center, Seoul
  - Seoul St.Mary Hospital, div hemato-oncology, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (12):
  - Institut Català D'Oncologia (ICO), Badalona, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres, Extremadura
  - Hosp.Universitario A Coruña-Hospital Teresa Herrera, A Coruña, Galicia
  - Hospital Universitario Son Espases, Palma de Mallorca, Isla Baleares
  - "Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Univers itario HM Sanchinarro, Madrid
  - Hospital Uni vcrsitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario y Politecnico de La Fe, Valencia
- Taiwan (7):
  - Changhua Christian Hospital, Changhua
  - Hematology and Oncology, Changhwa Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospita, Taichung
  - Division of Hematology, National Taiwan University Hospital, Taipei
  - koo-Foundation Sun Yat-Sen Cancer Center, Taipei
- United Kingdom (5):
  - Royal Devon & Exeter Hospital (Wonford site), Exeter, Devon
  - Blackpool Teaching Hospitals NHS Foundation Trust, Blackpool, Lancashire
  - Bradford Teaching Hospitals NHS Foundation trust, Bradford
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Royal Liverpool University Hospital, Liverpool

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Approx. 130 sites worldwide (planned), 116 sites where patients were randomized. Date of 1st patient screened: 12 Jul 2017 and Date of last patient completed: 08 Aug 2020
  A total of 725 patients were screened. Of these, 319 were considered screening failures, so a total of 406 patients were randomized
Pre-assignment Details: Based on request of the IDMC, the interim analysis was actually done on 30Jun2020 when 232/390 events occurred in the study, The study was stopped for futility.
Period: Overall Study
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Started | 203 (Screened patients) | 203 (Screened patients)
Treated | 201 | 201
Completed | 0 | 0
Not Completed | 203 | 203
Not completed — Adverse Event | 24 | 23
Not completed — Death | 46 | 26
Not completed — Physician Decision | 13 | 19
Not completed — Withdrawal by Subject | 16 | 20
Not completed — Progressive disease | 45 | 61
Not completed — non-compliance by patient | 1 | 0
Not completed — other reasons | 56 | 52
Not completed — randomized and not treated | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA | Total
Number analyzed (Participants) | 203 | 203 | 406
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 196 | 198 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.4 (5.48) | 75.1 (5.91) | 75.3 (5.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 87 | 174
  Male | 116 | 116 | 232
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 27 | 26 | 53
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 4 | 6
  White | 149 | 140 | 289
  More than one race | 3 | 3 | 6
  Unknown or Not Reported | 22 | 28 | 50
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 34 | 29 | 63
  Argentina | 3 | 2 | 5
  Brazil | 10 | 15 | 25
  Czechia | 10 | 8 | 18
  France | 8 | 10 | 18
  Germany | 5 | 6 | 11
  Hungary | 12 | 14 | 26
  Italy | 19 | 11 | 30
  Poland | 21 | 13 | 34
  South Korea | 8 | 7 | 15
  Romania | 10 | 7 | 17
  Spain | 24 | 28 | 52
  Taiwan | 17 | 18 | 35
  United Kingdom | 6 | 11 | 17
  United States | 12 | 18 | 30
  Austria | 4 | 6 | 10
Height [Mean (Standard Deviation); unit: cm] | 165.1 (10.23) | 165.7 (8.96) | 165.4 (9.61)
Smoking Habits [Count of Participants; unit: Participants]
  Non-smoker | 130 | 121 | 251
  Ex-smoker | 73 | 79 | 152
  Current smoker | 0 | 3 | 3
Cytogenetic Risk Category (central Lab results) [Count of Participants; unit: Participants] — Favorable: inv(16)/t(16;16)/del(16q), t(15;17) with/without secondary aberrations; t(8;21) lacking del (9q) or lacking complex karyotypes.
  Intermediate: Normal, +8, +6, -Y, del(12p)
  Unfavorable: del(5q)/-5, -7/del(7q), abn 3q, 9q, 11q, 20q, 21q, 17p, t(6;9), t(9;22) and complex karyotypes (≥ 3 unrelated abnormalities)
  Unknown: All other abnormalities
  Participants
    Intermediate | 109 | 107 | 216
    Unfavorable | 51 | 60 | 111
    Missing | 43 | 36 | 79
Cytogenetic Risk Category (local or central Lab results used for randomization) [Count of Participants; unit: Participants] — Favorable: inv(16)/t(16;16)/del(16q), t(15;17) with/without secondary aberrations; t(8;21) lacking del (9q) or lacking complex karyotypes.
  Intermediate: Normal, +8, +6, -Y, del(12p)
  Unfavorable: del(5q)/-5, -7/del(7q), abn 3q, 9q, 11q, 20q, 21q, 17p, t(6;9), t(9;22) and complex karyotypes (≥ 3 unrelated abnormalities)
  Unknown: All other abnormalities
  Participants
    Intermediate | 136 | 135 | 271
    unfavorable | 67 | 68 | 135
ECOG PS (used for randomization) [Count of Participants; unit: Participants] — Grade and Descriptions
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1. - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  2. - Ambulatory and capable of all selfcare, but unable to carry out any work activities; and about more than 50% of waking hours.
  3. - Capable of only limited self-care; confined to bed or chair more than 50% of waking hours.
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. - Dead
  Participants
    Grade 0-1 | 113 | 114 | 227
    Grade 2 | 90 | 89 | 179
ECOG PS (at cycle 1 Day 1) [Count of Participants; unit: Participants] — Grade and Descriptions
  0 - Fully active, able to carry on all pre-disease performance without restriction.
  1. - Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work).
  2. - Ambulatory and capable of all selfcare, but unable to carry out any work activities; and about more than 50% of waking hours.
  3. - Capable of only limited self-care; confined to bed or chair more than 50% of waking hours.
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. - Dead
  Participants
    Grade 0-1 | 114 | 110 | 224
    Grade 2 | 85 | 88 | 173
    Grade 3 | 0 | 1 | 1
    Missing | 4 | 4 | 8
Renal impairment [Count of Participants; unit: Participants]
  Normal or high: ≥ 90 mL/mg/1.73 m2 | 24 | 28 | 52
  Mildly decreased: 60-89 mL/mg/1.73 m2 | 118 | 102 | 220
  Mildly to moderately decreased: 45-59 mL/mg/1.73 m2 | 39 | 41 | 80
  Moderately to severely decreased: 30-44 mL/mg/1.73 m2 | 18 | 28 | 46
  Severely decreased: 15-29 mL/mg/1.73 m2 | 1 | 1 | 2
  Missing | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: OS measures the time from randomization to death due to any cause.
Time Frame: 826 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
days | 303 [209 to 400] | 303 [248 to 346]
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Superiority; p = 0.8275, Log Rank — P-value stratified by cytogenetic risk factor and ECOG performance status

2. Secondary Outcome: Morphologic Complete Remission (CR) Rate
Description: The CR rate is the proportion of patients who achieve a morphologic CR according to the response criteria
  * <5% blasts in a bone marrow aspirate sample with spicules
  * There should be no blasts with Auer rods
  * No EMD
  * Absolute Neutrophil Count (ANC) ≥1,000/μL
  * Platelet count of ≥100,000/μL
  * Patient must be independent of transfusions (for at least 1week before each assessment)
Time Frame: 744 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
Participants | 24 | 35
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.1244, Cochran-Mantel-Haenszel

3. Secondary Outcome: Complete Remission Without Minimal Residual Disease (CRmrd) Rate
Description: proportion of patients who achieve a CR without minimal residual disease by multicolor flow cytometry according to the following criteria
  * Morphologic CR
  * Minimal Residual Disease (MRD) by MFC negative
Time Frame: 826 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
Participants | 12 | 20
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.1430, Cochran-Mantel-Haenszel

4. Secondary Outcome: Cytogenetic Complete Remission (CRc) Rate
Description: The CRc rate is the proportion of patients who achieve a reversion to a normal karyotype at CR within the study period. This endpoint applies only to patients with abnormal cytogenetic at enrollment according to the following criterion
  Morphologic CR plus reversion to a normal karyotype (defined as no clonal abnormalities detected in a minimum of 20 mitotic cells)
Time Frame: 826 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 80 | 64
Participants | 7 | 8
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Superiority; p = 0.9977, Cochran-Mantel-Haenszel

5. Secondary Outcome: Transfusion Independence (TI)
Description: Transfusion independence rate is defined as the proportion of patients who show eight weeks or over without red blood cell (RBC-TI) and/or platelet (PLT-TI) transfusion during study period
Time Frame: 826 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
Participants | 81 | 81
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.9959, Cochran-Mantel-Haenszel

6. Other Pre Specified Outcome: Composite Complete Remission (cCR) Rate
Description: Composite complete remission (cCR) rate is the proportion of patients who achieve either a disease response of CR, CRi or MLFS (i.e., cCR = CR + CRi + MLFS) within the study period, according to the response criteria
Time Frame: 744 days
Measure: Count of Participants; unit: Participants
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
Participants | 73 | 64
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.3502, Cochran-Mantel-Haenszel

7. Other Pre Specified Outcome: Duration of Composite Complete Remission
Description: Duration of cCR response is the time from first cCR until documented relapse (the definition of relapse from CR will be applied) or death. Duration of cCR is only defined for patients who achieve a cCR
Time Frame: 744 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 73 | 64
days | 576 [276 to NA] — The upper confidence limit for median cannot be estimated (and it was reported as NA) as the curve that represents the upper confidence limits for the survivor function lies above 0.50. The LogLog transformation was used for computing the confidence interval | 319 [170 to 744]
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.0502, Log Rank

8. Other Pre Specified Outcome: Change in Quality of Life From Baseline (EORTC QLQ-C30 - European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30)
Description: QLQ-C30 is made of multi-item scales and single-item measures (functional and symptom scales, a global health status/QoL scale and single items). Item range is the difference between possible max and min response to individual items of the scale; most items take values from 1 to 4 (range=3). Global health status takes values from 1 to 7 (range = 6). For statistical analysis purpose, single-item and scale values were all standardized (according to linear transformation described in Scoring Manual) to obtain scores ranging 0-100. An high scale score represents an higher response level. Thus an high score for a functional scale represents an high/healthy level of functioning, an high score for the global health status/QoL represents a high QoL, an high score for a symptom scale/item represents an high level of symptomatology/problems.
Time Frame: from baseline up to 660 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
score on a scale
  Global Health Status | -7.040 (31.4458) | -2.303 (28.6611)
  Functional Scale - Physical Functioning | -8.937 (32.1163) | -7.018 (25.8512)
  Functional Scale - Role Functioning | -6.034 (46.3793) | -2.000 (40.2659)
  Symptom Scale - Fatigue | 2.107 (34.2928) | 4.240 (29.7030)
  Symptom Scale - Nausea and Vomiting | 5.460 (28.1649) | 5.263 (23.2870)
  Symptom Scale - Appetite Loss | 9.771 (42.8107) | 3.509 (40.2150)

9. Other Pre Specified Outcome: Relapse Free Survival
Description: the time from the date of achievement of CR or CRi until the date of relapse or death from any cause
Time Frame: 744 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
days | 291 [217 to 429] | 190 [155 to 319]
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.4656, Log Rank

10. Other Pre Specified Outcome: Progressive Free Survival Rate (PFS)
Description: PFS is defined as the time from the date of randomization until the date of relapse (progression), or death from any cause, whichever occurs first.
Time Frame: 800 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
days | 217 [126 to 257] | 220 [182 to 271]
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.7063, Log Rank

11. Other Pre Specified Outcome: Duration of Morphologic CR
Description: Duration of morphologic CR is defined as the time from the date of achievement of CR until the date of relapse (progression).
Time Frame: 744 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 24 | 35
days | NA [352 to NA] — Median was not reachable due to low number of patients with events (CR) therefore the upper limit is not computable | 319 [119 to 744]
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.0592, Log Rank

12. Other Pre Specified Outcome: Time to CR
Description: Time to CR is defined as the time from the date of randomization until the date of CR in the absence of interceding therapies. The analysis set was the ITT set.
Time Frame: 616 days
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
days | NA [NA to NA] — Time to CR was censored at the date of the last assessment of patient status excluding CR in case no CR occurred by time of analysis. The number of subjects reaching CR was lower than 50%, then neither the median nor the confidence interval were computable | 361 [311 to NA] — The upper confidence limit for median cannot be estimated (and it was reported as NA) as the curve that represents the upper confidence limits for the survivor function lies above 0.50. The LogLog transformation was used for computing the confidence interval
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.3835, Log Rank

13. Other Pre Specified Outcome: Morphologic CR Within 6 Cycles Rate
Description: Morphologic CR within 6 cycles rate is defined as the proportion of patients who achieved CR in the absence of interceding therapies within 6 treatment cycles (i.e., during treatment phase up to Day 1 of Cycle 7 included). Analysis was performed in the ITT set.
Time Frame: within 6 cycles
Measure: Number; unit: number of patients
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
Number analyzed (Participants) | 203 | 203
number of patients | 14 | 16
Statistical Analysis 1: Comparison: Pracinostat Plus AZA vs Placebo Plus AZA; Test type: Other; p = 0.7099, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: TEAEs are with onset date/time at or after start date/time of first intake of pracinostat /placebo, or AEs with onset date/time prior to start date/time of first intake of pracinostat/placebo that worsen in severity after start date/time of first intake of pracinostat /placebo, up to end of observation period. Observation period is defined as 30 days after last dose of pracinostat/placebo or start of new therapy for AML whichever occurs first up to 672 days. OS was collected up to 826 days.
Description: When evaluating all-cause mortality, the population at risk included all the patients randomized (203 patients per each arm) being the mortality linked to the efficacy endpoint.
  When evaluating Adverse Events, the population at risk included patients who received at least one dose of treatment (201 patients per each arm).
Arm/Group | Pracinostat Plus AZA | Placebo Plus AZA
All-Cause Mortality (participants affected / at risk) | 121/203 | 128/203
Serious Adverse Events (participants affected / at risk) | 153/201 | 151/201
Other Adverse Events (participants affected / at risk) | 197/201 | 193/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pracinostat Plus AZA (N=201) | Placebo Plus AZA (N=201)
Pneumonia (Infections and infestations) | 25 (27) | 31 (37)
Sepsis (Infections and infestations) | 18 (20) | 15 (17)
Urinary tract infection (Infections and infestations) | 9 (16) | 6 (6)
Cellulitis (Infections and infestations) | 5 (5) | 5 (5)
Septic shock (Infections and infestations) | 5 (5) | 4 (4)
Lung infection (Infections and infestations) | 5 (5) | 3 (3)
Bacteraemia (Infections and infestations) | 5 (6) | 2 (2)
Neutropenic sepsis (Infections and infestations) | 4 (6) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 60 (105) | 53 (79)
Anaemia (Blood and lymphatic system disorders) | 9 (11) | 9 (16)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (8) | 5 (10)
Pancytopenia (Blood and lymphatic system disorders) | 5 (10) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Pyrexia (General disorders) | 11 (12) | 15 (17)
Fatigue (General disorders) | 6 (7) | 2 (2)
Vomiting (Gastrointestinal disorders) | 7 (7) | 2 (2)
Nausea (Gastrointestinal disorders) | 6 (6) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (9) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 5 (6) | 2 (2)
Nervous system disorders (Nervous system disorders) | 10 (11) | 9 (10)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 10 (12) | 5 (5)
Vascular disorders (Vascular disorders) | 8 (8) | 5 (7)
Investigations (Investigations) | 8 (9) | 3 (3)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3) | 6 (7)
Renal and urinary disorders (Renal and urinary disorders) | 3 (3) | 6 (6)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (7)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pracinostat Plus AZA (N=201) | Placebo Plus AZA (N=201)
Nausea (Gastrointestinal disorders) | 85 (125) | 79 (101)
Vomiting (Gastrointestinal disorders) | 64 (96) | 50 (80)
Constipation (Gastrointestinal disorders) | 56 (76) | 60 (76)
Diarrhoea (Gastrointestinal disorders) | 54 (83) | 35 (52)
Anaemia (Blood and lymphatic system disorders) | 59 (126) | 69 (158)
Febrile neutropenia (Blood and lymphatic system disorders) | 69 (123) | 61 (97)
Thrombocytopenia (Blood and lymphatic system disorders) | 44 (97) | 41 (88)
Neutropenia (Blood and lymphatic system disorders) | 37 (63) | 32 (68)
Pneumonia (Infections and infestations) | 36 (39) | 44 (54)
Pyrexia (General disorders) | 43 (68) | 45 (76)
Fatigue (General disorders) | 37 (44) | 38 (48)
Hypokalaemia (Metabolism and nutrition disorders) | 48 (80) | 39 (60)
Decreased appetite (Metabolism and nutrition disorders) | 39 (52) | 31 (35)
Investigations (Investigations) | 74 (223) | 60 (108)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 73 (138) | 85 (159)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 56 (89) | 57 (100)
Nervous system disorders (Nervous system disorders) | 61 (88) | 62 (84)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 41 (79) | 59 (86)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 36 (65) | 46 (62)
Vascular disorders (Vascular disorders) | 54 (72) | 39 (50)
Cardiac disorders (Cardiac disorders) | 41 (59) | 39 (58)
Renal and urinary disorders (Renal and urinary disorders) | 32 (46) | 50 (68)
Psychiatric disorders (Psychiatric disorders) | 35 (47) | 40 (47)
Abdominal pain (Gastrointestinal disorders) | 16 (18) | 15 (17)
Haemorrhoids (Gastrointestinal disorders) | 16 (18) | 11 (13)
Proctalgia (Gastrointestinal disorders) | 10 (12) | 6 (7)
Mouth ulceration (Gastrointestinal disorders) | 12 (13) | 5 (5)
Urinary tract infection (Infections and infestations) | 21 (29) | 18 (23)
Sepsis (Infections and infestations) | 18 (20) | 15 (17)
Upper respiratory tract infection (Infections and infestations) | 17 (19) | 7 (8)
Oral candidiasis (Gastrointestinal disorders) | 11 (13) | 11 (11)
Oedema peripheral (General disorders) | 29 (42) | 31 (37)
Asthenia (General disorders) | 24 (32) | 17 (19)
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 (23) | 19 (38)
Hypophosphataemia (Metabolism and nutrition disorders) | 17 (18) | 9 (10)
Hyperglycaemia (Metabolism and nutrition disorders) | 12 (12) | 11 (11)
Hyponatraemia (Metabolism and nutrition disorders) | 10 (12) | 7 (8)
Platelet count decreased (Investigations) | 23 (69) | 7 (8)
Neutrophil count decreased (Investigations) | 16 (46) | 13 (18)
Weight decreased (Investigations) | 24 (26) | 15 (15)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 15 (18) | 28 (29)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (20) | 20 (23)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 (9) | 13 (13)
Rash (Skin and subcutaneous tissue disorders) | 12 (14) | 10 (11)
Dizziness (Nervous system disorders) | 13 (14) | 22 (26)
Headache (Nervous system disorders) | 14 (20) | 12 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (17) | 23 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 12 (12) | 9 (9)
Transfusion reaction (Injury, poisoning and procedural complications) | 10 (20) | 4 (6)
Fall (Injury, poisoning and procedural complications) | 10 (12) | 6 (6)
Hypertension (Vascular disorders) | 13 (14) | 15 (18)
Hypotension (Vascular disorders) | 17 (20) | 11 (11)
Haematoma (Vascular disorders) | 10 (10) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 17 (23) | 13 (16)
Acute kidney injury (Renal and urinary disorders) | 13 (13) | 12 (14)
Insomnia (Psychiatric disorders) | 15 (18) | 7 (9)

LIMITATIONS AND CAVEATS:
Results of the interim analysis (OS curves crossing at about 300 days) demonstrated futility according to the planned threshold and concluded that it was unlikely to meet the primary endpoint compared to the control group at the final analysis. Based on this outcome, the decision taken was to discontinue the recruitment of patients and terminate the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT03151408/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-11): https://cdn.clinicaltrials.gov/large-docs/08/NCT03151408/SAP_001.pdf